CLINICAL TRIAL: NCT06817109
Title: Implementation of Internet-based Psychotherapy for Symptoms of Depression, Insomnia and Anxiety in Primary Care in the Cities of Indaiatuba and Jaguariuna
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81434224.9.0000.0068
Record Dates: First submitted 2024-08-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Depression; Insomnia; Anxiety
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: comparison between the intervention and the treatment as usual
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iCBT (Experimental): For participants allocated to ICBT, in addition to the usual care performed in the primary unit, these individuals will also receive digital intervention through an online platform specifically developed for this purpose. Depression and anxiety intervention will consist of 10 specific modules for the treatment of each disorder to be performed within 10 weeks. Insomnia intervention will consist of 9 specific modules for the treatment of insomnia, to be performed within 8 weeks. These modules use concepts associated with cognitive behavioral therapy and third-generation behavioral therapy and were created through the transcultural and digital adaptation the therapeutic ingredients present in consumed treatment manuals in the literature.
  In all modules, a therapist will be designated to accompany each patient.
  Interventions: Device: interactive technological intervention for improvement of mental health symptoms in Primary Care users Health
- Treatment as usual (No Intervention): Patients allocated to this arm will continue to receive the usual treatment in their health units, which usually consists of psychotropic drugs and psychological support

INTERVENTIONS:
Device: interactive technological intervention for improvement of mental health symptoms in Primary Care users Health — Intervention based on cognitive and behavioral techniques, such as psychoeducation on anxiety, depression and insomnia; muscle relaxation and breathing techniques; sleep hygiene techniques, behavioral activation and mindfulness techniques
  Other Names: CONEMO
  Arms: iCBT

SUMMARY:
The main objective of this study is to evaluate the effectiveness and success of implementing internet-based cognitive behavioral psychotherapy (iCBT) guided by a therapist for symptoms of depression, insomnia and anxiety in individuals who did not respond to an automated intervention in primary care in the cities of Indaiatuba and Jaguariúna. Method: This is a pragmatic, prospective, randomized, two-arm, parallel-group, controlled clinical trial, comparing a therapist-guided Internet-based cognitive behavioral therapy (iCBT) treatment associated with usual care versus usual care alone (UC) for symptoms of depression, insomnia and anxiety in adults who attend primary care in the cities of Indaiatuba and Jaguariúna and who did not respond to a first phase of treatment with automated iCBT (not guided by a therapist) focused on these groups of symptoms. The results will be accessed during treatment, in the immediate post-treatment (after two weeks of completing treatment) and at 3 and 6 month follow-up.

DETAILED DESCRIPTION:
Hypotheses:

Guided iCBT will produce an additive effect of significant reduction in symptoms of depression, insomnia, and anxiety compared to treatment as usual.

Design Plan:

Study type Experiment - A researcher randomly assigns treatments to study subjects, this includes field or lab experiments. This is also known as an intervention experiment and includes randomized controlled trials.

Blinding Personnel who analyze the data collected from the study are not aware of the treatment applied to any given group.

Study design This is a pragmatic, prospective, randomized, two-arm, parallel-group, controlled clinical trial, comparing a therapist-guided Internet-based cognitive behavioral therapy (iCBT) treatment associated with usual care versus usual care alone (UC) for symptoms of depression, insomnia and anxiety in adults who attend primary care in the cities of Indaiatuba and Jaguariúna and who did not respond to a first phase of treatment with automated iCBT (not guided by a therapist) focused on these groups of symptoms. The results will be accessed during treatment, in the immediate post-treatment (after two weeks of completing treatment) and at 3 and 6 month follow-up.

Randomization The patient will be randomized to receive or not receive the iCBT intervention in addition to their usual treatment in a 1:1 ratio. Randomization will be electronic and carried out by software, and will use stratification techniques by sex, severity of the underlying disorder, use of psychiatric medication, socioeconomic level, and age. Participants will be randomized between iCBT groups specific to their primary disorder in addition to usual treatment, or only the Usual care (UC) provided in a Basic Health Unit (including psychosocial counseling, drug treatment, or others available in the public network).

Sampling Plan

Existing Data Registration prior to analysis of the data

Data collection procedures This is the second phase of a study that will recruit participants in the 28 Basic Health Units in the municipalities of Indaiatuba and Jaguariúna. In this second phase, individuals will be included who, after receiving a completely automated intervention via a cell phone application for symptoms of Depression, Anxiety and Insomnia (CONEMO), persist with significant complaints and are motivated to participate in more intensive treatment.

Adults aged between 18 and 65 will be eligible, who have access to the internet and who participated in the first phase of a study that will use CONEMO which provides for the provision of cognitive behavioral intervention for treating symptoms of depression, insomnia and anxiety using an app.

At the end of application treatment in the first phase of the study, patients who persist with high levels of Depression (PHQ-9 >= 10), Insomnia (IGI >= 11) or Anxiety (GAD-7) will receive a link to access a initial electronic first screening form, hosted on a digital platform. The possibility of questioning a representative of the research group will be ensured if they do not understand the question asked or refuse to answer if the participant does not feel comfortable doing so. To minimize the risk of breach of privacy and confidentiality, we will use a secure server to store data, protected by a password and accessed from secure computers.

Individuals who meet inclusion criteria will be assessed by a trained clinical psychologist in an online session, where the primary diagnosis will be confirmed by structured clinical interview. The patient will be randomized to receive or not receive the iCBT intervention in addition to their usual treatment in a 1:1 ratio. It is important to mention that confirmation or not of the main diagnosis is not an inclusion or exclusion criterion, which are based on dimensional scales of symptoms, but will be used in effectiveness subgroup analyzes (i.e., to verify whether the formal clinical diagnosis is associated to a more significant response due to greater precision of the associated treatment). Randomization will be electronic and carried out by software, and will use stratification techniques by sex, severity of the underlying disorder, use of psychiatric medication, socioeconomic level, and age. Participants will be randomized between iCBT groups specific to their primary disorder in addition to usual treatment, or only the Usual Treatment/Care (UC) provided in a Basic Health Unit (including psychosocial counseling, drug treatment, or others available in the public network).

Sample size Our target sample size is 232 participants. We will attempt to recruit up to 268, assuming 15% of attrition rate.

Sample size rationale Based on estimates from the study by Araya, Menezes, Claro et al (2021), G-Power was used to calculate the total sample size necessary to detect an odds ratio (OR) of 1.4 difference between responders and non-responders to the treatment for depression, insomnia and anxiety (50% reduction in PHQ-9 and/or GAD-7 and/or 8 point reduction in ISI) between groups (ITCC vs TU). This difference of 1.4 comes from the comparison of responders and non-responders (41% vs 29%) in the study by Araya, Menezes, Claro et al (2021). Using the logistic regression test, G-Power indicated a sample size of 268 (232 + 36 attrition rate) considering a 5% significance level, 80% power and 15% attrition rate.

Variables Manipulated variables For participants allocated to iCBT, in addition to the usual care provided in the primary unit, these individuals will also receive digital intervention through an online platform specifically developed for this purpose. The depression and anxiety intervention will consist of 10 specific modules for the treatment of each disorder, to be carried out over a period of 10 weeks. The insomnia intervention will consist of 9 modules specific to the treatment of insomnia, to be carried out over a period of 8 weeks. These modules use concepts associated with Cognitive-Behavioral Therapy and Contextual Behavioral Therapy and were created through cross-cultural adaptation and for the digital environment the therapeutic ingredients present in treatment manuals recognized in the literature. The researchers involved in this adaptation are therapists experienced in applying these protocols and conducting clinical psychotherapy studies using these concepts. These researchers will also be responsible for training and supervising therapists from the city itself who will provide assistance to patients in the study.

In all modules, a therapist will be assigned to monitor each patient. All communication between patient and therapist will be carried out and stored on the platform (through electronic messages). The therapist will monitor the patient's progress, offer guidance and feedback throughout sessions, and answer questions the patient may have. In the iCBT protocol, participants will receive usual care in the primary unit plus the protocol for each disorder. All protocols were developed based on the theoretical framework of Cognitive Behavioral Therapy (CBT) and based on specific protocols for depression (PERINI et al., 2009), insomnia (HARVEY et al., 2014; EL RAFIHI-FERREIRA et al., 2020) and anxiety (FARCHIONE et al., 2012; ROY-BYRNE et al., 2010; BRASIL, 2021; Salum et al., 2020) which were effective in previous studies.

Measured variables Effectiveness outcomes will be compared between participants who received guided iCBT treatment in addition to treatment as usual and participants who only received treatment as usual.

Primary outcome:

Response to treatment for common emotional symptoms, which is a combined outcome defined by a significant reduction in symptoms of the disorder for the treatment to which the patient was allocated:

Depressive symptoms: Reduction of 50% or more in PHQ-9 score at 3-month follow-up.

Insomnia symptoms: Reduction of 8 points or more in the ISI score at 3-month follow-up Anxiety Symptoms: Reduction of at least 50% in the GAD-7 score at 3-month follow-up.

Secondary outcomes:

Response to treatment for common emotional symptoms at post-treatment (2 weeks after completing treatment) and at 6-month follow-up.

Remission of common emotional symptoms, which is a composite outcome defined by a final scale below that considered clinically significant (i.e., final score of less than 10 points on the PHQ-9 depression scale, final score of less than 8 points on the ISI insomnia scale , and a final score of less than 10 points on the GAD-7 Anxiety scale) in post-treatment and 3 and 6 month follow-up.

Linear (continuous) reduction in the total score of the PHQ-9 scale in post-treatment and 3 and 6 month follow-up.

Linear (continuous) reduction in the total IGI scale score in post-treatment and 3 and 6 month follow-up.

Linear (continuous) reduction in the total score of the I GAD-7 scale in post-treatment and 3 and 6 month follow-up.

Quality of life assessment: Linear evolution of the total score and sub-scores of the 12-Item Short-Form Health Survey (SF-12) scale: Total score; Physical domain score; Mental domain score in post-treatment and 3 and 6 month follow-up.

Sleep patterns assessed by the sleep diary: Sleep onset latency, night waking duration, total sleep time and sleep efficiency (relationship between sleep time and time spent in bed) post-treatment.

Analysis Plan Statistical models To measure the primary outcome, that is, response (success) to treatment, binary variables will be used to show whether the participant achieved a response (PHQ-9_3months - PHQ-9pre ≥50%; GAD-7_3months - GAD-7pre ≥50%; ISI_3months - ISIpre ≥ 8). These variables will be used as results of logistic regression models, where group fixed effects (iCBT vs. UT) will be included as predictors.

Logistic regression will also be used for categorical secondary outcomes such as post-treatment remission (PHQ-9 < 10; GAD-7 < 10; ISI < 8) and maintenance of response and remission at three and six month follow-up.

For secondary outcomes of continuous variables tests using Generalized Estimated Equations (GEE) or General Mixed Models (GMM) will be used to compare groups (iCBT versus UT) on changes in outcome variables over time (baseline, treatment, post-treatment and follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Participants included in the first phase of the study;
* Depression complaints with significant scores for depression> = 10 points; and/or
* Insomnia complaints with significant score for insomnia> = 11; and/or
* Complaints of significant score for anxiety> = 10.
* participants with significant symptoms in more than one domain, together with the professional, will be invited to elect a main focus of treatment, or by be the main problem and/or the one the patient is most motivated to treat.

Exclusion Criteria:

* Individuals who have acute suicide risk, evaluated by positive response (1, 2 or 3) to PHQ-9 item 9 and considered severe (suicidal illusion) in the Suicide Risk Assessment Protocol (S-RAP) will be excluded.
* Individuals identified as bass in S-rap will be sent for emergency care according to security monitoring protocol presented in the topic "Evaluation and Risk Monitoring" of this project.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 - Patient Health Questionnaire-9 | 3 month follow up
  Reduction of 50% or more in the PHQ-9 score
ISI - Insomnia Severity Index | 3 month follow up
  Reduction of 8 points or more in the ISI score
GAD-7 - Generalized Anxiety Disorder 7-item | 3 month follow up
  Reduction of 50% or more in the GAD-7

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Rossi Menezes, PhD, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Basic Health System, Indaiatuba, São Paulo
  - Basic Health System, Jaguariúna, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Data and analysis codes will be shared on the OSF platform after the study is published and under request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the studies are published.
Access Criteria: Upon request from others researchers.